CLINICAL TRIAL: NCT01594528
Title: Behavior During Experimentally Induced Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Dominique Malauzat, MD, Head of Research Department, Centre Hospitalier Esquirol
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-A00048-35
Record Dates: First submitted 2012-03-13; First posted 2012-05-09 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Schizophrenia; Major Depression
Keywords: schizophrenia; major depression; pain; behavior
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Pain; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SC (Experimental): behavior as defined with facial, corporal and vocal indicators during experimental pain tests for subjects with schizophrenia
  Interventions: Other: pain tests
- controls (Experimental): behavior as defined with facial, corporal and vocal indicators during experimental pain tests for subjects without any psychiatric trouble
  Interventions: Other: pain tests
- MD (Experimental): behavior as defined with facial, corporal and vocal indicators during experimental pain tests for subjects with major depression
  Interventions: Other: pain tests

INTERVENTIONS:
Other: pain tests — pain induction with pressure application or ischemia on the arm

SUMMARY:
Numerous factors can influence the processing of pain message: the affective or emotional, the sensorial and the cognitive components. Interindividual variations at the emotional and cognitive levels may interfere with the pain message and the consecutive behavior. Some modifications in these components are observed in psychiatric troubles, but their influences on the behavior to pain have not been studied, although they have been studied in some populations characterized as non communicating, with obvious cognitive degradations (subject with dementia, older, newborns,…).In an other study in course, the past pain experience is explored in relation to results to experimental pain tests, emotional and anxious characteristics. This present pilot study aims at studying the infra-verbal behavioural signs during experimentally induced pain in subjects with schizophrenia, major depression, and controls.

DETAILED DESCRIPTION:
The objective is to search for behavioral non verbal indicators of pain during experimentally induced pain (pressure application, ischemia induction).

Included subjects are subjected to experimental pain tests : pressure application (160 kPa) with an algometer to determine the pain with Visual Analogic Scale (VAS), and ischemia induction to determine the time needed to feel pain with an intensity equivalent to 3 with the VAS.

Subjects are filmed during experimentation to identify the corporal mobility signs, facial expression signs and sonorous signs associated to pain stimulation.

Neurophysiological measures complete these observations : surface electromyogram, heart rate measure, blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* subjects with psychiatric trouble : diagnosis of schizophrenia or major depression according to the DSM-IV-TR criteria.
* control subjects : without known psychiatric history.
* age between 18 and 60.

Exclusion Criteria:

* absence of consent, hospitalization under constraint, absence of health insurance.
* inability to answer the questionnaires
* pregnancy
* antalgic or analgesic treatment
* allergy to latex
* non stabilized high blood pressure, bad blood coagulation,
* peripheral neuropathy, nerve lesion, dermatosis at the superior extremities, muscular lesion or pathology at the upper member level
* non treated alcohol dependence
* illegal substance consumption in the past 48 hours
* participation to an other biomedical study during the 2 weeks before inclusion, and until the pain tests, if this study can interfere with the realization of the objectives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Malauzat, MD, Principal Investigator — Centre Hospitalier Esquirol
Locations (1):
- Centre Hospitalier Esquirol, Limoges, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: behavior during experimental pain tests for control subjects
  pain tests: pain induction with pressure application or ischemia on the arm
- SChizophrenia: behavior during experimental pain tests for subjects with schizophrenia
  pain tests: pain induction with pressure application or ischemia on the arm
- Major Depression: behavior during experimental pain tests for subjects with major depression pain tests: pain induction with pressure application or ischemia on the arm
Period: Overall Study
Arm/Group | Control | SChizophrenia | Major Depression
Started | 16 | 17 | 16
Completed | 16 | 17 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: subjects with major depression
Groups:
- Major Depression: subjects with major depression
- Schizophrenia: subjects with schizophrenia
- Control: subjects without psychiatric disorders
- Total: Total of all reporting groups
Arm/Group | Major Depression | Schizophrenia | Control | Total
Number analyzed (Participants) | 16 | 17 | 16 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [37.5 to 51.5] | 42 [35 to 49] | 40 [33.5 to 48.5] | 41 [35 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 6 | 22
  Male | 3 | 14 | 10 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  France | 16 | 17 | 16 | 49

OUTCOME MEASURES:

1. Primary Outcome: Indicators / Minute
Description: number of corporal mobility, facial expression and sound indicators
Time Frame: during pain tests (average 1 hour)
Measure: Median (95% Confidence Interval); unit: indicators/minute
Groups:
- Group of Subjects Presenting Schizophrenia SC: subjects with diagnosis of schizophrenia according to the DSM-IV-TR and experimentating pain tests: pain induction with pressure application or ischemia on the arm.
  and observation of the behavior as defined with facial, corporal and vocal indicators during experimental pain tests
- Group of Subjects Presenting Major Depression MD: subjects presenting a diagnosis of major depression according to the DSM-IV-TR and experimentating pain tests: pain induction with pressure application or ischemia on the arm.
  and observation of the behavior as defined with facial, corporal and vocal indicators during experimental pain tests
- Group of Subjects Without Psychiatric Troubles C: control subjects without any psychiatric disorder and experimentating the same pain tests as the other groups: pain induction with pressure application or ischemia on the arm.
  and observation of the behavior as defined with facial, corporal and vocal indicators during experimental pain tests
Arm/Group | Group of Subjects Presenting Schizophrenia SC | Group of Subjects Presenting Major Depression MD | Group of Subjects Without Psychiatric Troubles C
Number analyzed (Participants) | 17 | 16 | 16
indicators/minute
  vocal indicators | 1.925 [0 to 2.4] | 0.23 [0 to 4.23] | 0.4 [0 to 1.15]
  body indicators | 0.45 [0 to 1.6] | 0.59 [0 to 2.1] | 0.55 [0 to 2.7]
  facial indicators | 0.25 [0 to 1.5] | 0.4975 [0.1 to 3.95] | 0.45 [0.1 to 4.25]
Statistical Analysis 1: Comparison: Group of Subjects Presenting Schizophrenia SC vs Group of Subjects Presenting Major Depression MD vs Group of Subjects Without Psychiatric Troubles C; Test type: Other; p = 0.992, Wilcoxon (Mann-Whitney) — comparison between groups for body indicators
Statistical Analysis 2: Comparison: Group of Subjects Presenting Schizophrenia SC vs Group of Subjects Presenting Major Depression MD vs Group of Subjects Without Psychiatric Troubles C; Test type: Other; p = 0.8, Wilcoxon (Mann-Whitney) — comparison between groups facial indicators
Statistical Analysis 3: Comparison: Group of Subjects Presenting Schizophrenia SC vs Group of Subjects Presenting Major Depression MD vs Group of Subjects Without Psychiatric Troubles C; Test type: Other; p = 0.586, Wilcoxon (Mann-Whitney) — comparison between groups for vocal indicators

ADVERSE EVENTS:
Time Frame: 12 months
Description: no adverse event to be reported
Groups:
- Diagnosis: diagnosis according to the DSM-IV-TR : major depression and schizophrenia, or control.
  pain tests: pain induction with pressure application or ischemia on the arm
Arm/Group | Diagnosis
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes